CLINICAL TRIAL: NCT01483625
Title: A 12-week, Randomised, Placebo-controlled, Double-blind, Parallel Group, Multi-center Trial to Assess the Efficacy and Safety of Tiotropium Bromide (18 µg) Delivered Via the HandiHaler® in Patients With Newly Diagnosed and/or Maintenance Treatment naïve Chronic Obstructive Pulmonary Disease (COPD) Experiencing an Acute Respiratory Infection (TICARI 1: Tiotropium In COPD Patients With an Acute Respiratory Infection 1)
Brief Title: Tiotropium (18mcg) in Chronic Obstructive Pulmonary Disease (COPD) Patients With a Respiratory Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.479
Record Dates: First submitted 2011-11-30; First posted 2011-12-01 (Estimated); Results first posted 2014-04-10 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- tiotropium 18mcg (Experimental): active
  Interventions: Drug: tiotropium
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: tiotropium — 18mcg
  Arms: tiotropium 18mcg
Drug: Placebo — placebo
  Arms: Placebo

SUMMARY:
The aim of the study is to investigate whether the early introduction of maintenance bronchodilator therapy during an acute symptomatic episode of the disease shows benefits on the recovery of symptoms. It also represents an opportunity to identify COPD patients earlier in their disease state and start maintenance therapy, if appropriate.

ELIGIBILITY:
Inclusion criteria:

1. All patients must sign an informed consent consistent with International Conference on Harmonization - Good Clinical Practice (ICH-GCP) guidelines prior to participation in the trial and conducting any study procedures.
2. Male or female patients 40 years of age or older.
3. Ability to independently read and understand English and/or Spanish.
4. Any self-reported history of smoking (e.g. = 100 cigarettes (~5 packs) during life-time).
5. Acute respiratory symptoms for up to 7 days
6. All patients must have a diagnosis of COPD, and must have an airway obstruction with a post-bronchodilator (Forced Expiratory Volume in 1 second (FEV1)/Forced Vital Capacity (FVC)) <0.7. The diagnosis of COPD can be made at Visit 1.
7. The clinical assessment of the enrolled patient in the judgement of the investigator supports the introduction of COPD maintenance therapy.
8. Patients must be able to inhale medication in a competent manner from the HandiHaler® device and from a metered dose inhaler (MDI)

Exclusion criteria:

1. Therapy with any long-acting bronchodilator, short-acting anticholinergic, inhaled corticosteroid or regular maintenance use (>14 consecutive days) of systemic corticosteroid (the latter for respiratory indications) during the previous 6 months (short course of systemic corticosteroid for up to 14 days for respiratory indications allowed); in case of use of systemic corticosteroid medication for other than respiratory conditions, then exclusion of unstable doses (i.e., less than six weeks on stable dose) or at doses in excess of the equivalent of 10 mg prednisolone-equivalent per day. In addition, daily use of short-acting beta2-agonist for more than a week prior to Visit 0 not allowed.

   The following exclusion criteria apply at Visit 1:
2. Significant diseases other than COPD. A significant disease is defined as a disease or condition which, in the opinion of the investigator, may put the patient at risk because of participation in the study or may influence the patient¿s ability to participate in the study.
3. A recent history (i.e., six months or less) of myocardial infarction. Patients being stable with a history of cardiac stents prior to six month are permitted.
4. Any unstable or life-threatening cardiac arrhythmia requiring intervention or change in drug therapy during the last year.
5. Hospitalisation for cardiac failure (New York Heart Association (NYHA) Class III or IV) during the past year.
6. Any significant or new ECG findings at V1 as judged by the investigator, including, but not limited to signs of ischemia, arrhythmia, heart failure, or the report of chest pain.
7. Known active tuberculosis.
8. Current asthma (patient treated for asthma in the last 2 years), cystic fibrosis, clinical diagnosis of bronchiectasis, interstitial lung disease, or pulmonary thromboembolic disease.
9. A history of thoracotomy with pulmonary resection. Patients with a history of thoracotomy for other reasons should be evaluated as per exclusion criterion no. 2.
10. Malignancy for which the patient has undergone resection, radiation, chemotherapy or biological treatments within the last year or is currently on active radiation therapy, chemotherapy or biological treatment. Patients with treated basal cell carcinoma are allowed.
11. At visit 0 or 1, a severe respiratory infection, e.g. pneumonia (as suspected by investigator), any condition or exacerbation requiring ER visit or hospitalization, need for oxygen treatment.
12. Known hypersensitivity to anticholinergic drugs, lactose, or any other components of the HandiHaler® or MDI inhalation solution delivery system.
13. Treatment with any restricted pulmonary medication
14. Requirement of supplemental oxygen therapy for = 24 hours during the previous 6 months.
15. Known moderate to severe renal impairment.
16. Known narrow angle glaucoma.
17. Significant symptomatic prostatic hyperplasia or bladder-neck obstruction. Patients whose symptoms are controlled on treatment may be included.
18. Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception (i.e., oral contraceptives, intrauterine devices, diaphragm or subdermal implants e.g., Norplant®) for at least three months prior to and for the duration of the trial.
19. Significant alcohol or drug abuse within the past 12 months.
20. Actively participating in a pulmonary rehabilitation program.
21. Previously randomized in this study or currently participating in another interventional study.
22. Visual impairment that as judged by the investigator does not allow the patient to independently read and complete the questionnaires and electronic diary (eDiary).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2011-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (27):
- United States (27):
  - 205.479.01017 Boehringer Ingelheim Investigational Site, Tucson, Arizona
  - 205.479.01036 Boehringer Ingelheim Investigational Site, Riverside, California
  - 205.479.01024 Boehringer Ingelheim Investigational Site, San Diego, California
  - 205.479.01043 Boehringer Ingelheim Investigational Site, DeLand, Florida
  - 205.479.01040 Boehringer Ingelheim Investigational Site, St. Petersburg, Florida
  - 205.479.01022 Boehringer Ingelheim Investigational Site, Chelsea, Michigan
  - 205.479.01041 Boehringer Ingelheim Investigational Site, Picayune, Mississippi
  - 205.479.01037 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 205.479.01005 Boehringer Ingelheim Investigational Site, Tabor City, North Carolina
  - 205.479.01008 Boehringer Ingelheim Investigational Site, Wilmington, North Carolina
  - 205.479.01003 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 205.479.01002 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
  - 205.479.01044 Boehringer Ingelheim Investigational Site, Tipton, Pennsylvania
  - 205.479.01006 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 205.479.01001 Boehringer Ingelheim Investigational Site, Columbia, South Carolina
  - 205.479.01007 Boehringer Ingelheim Investigational Site, Easley, South Carolina
  - 205.479.01026 Boehringer Ingelheim Investigational Site, Fort Mill, South Carolina
  - 205.479.01031 Boehringer Ingelheim Investigational Site, Gaffney, South Carolina
  - 205.479.01012 Boehringer Ingelheim Investigational Site, Greenville, South Carolina
  - 205.479.01048 Boehringer Ingelheim Investigational Site, Hodges, South Carolina
  - 205.479.01004 Boehringer Ingelheim Investigational Site, Spartanburg, South Carolina
  - 205.479.01019 Boehringer Ingelheim Investigational Site, Union, South Carolina
  - 205.479.01039 Boehringer Ingelheim Investigational Site, Rapid City, South Dakota
  - 205.479.01033 Boehringer Ingelheim Investigational Site, Chattanooga, Tennessee
  - 205.479.01028 Boehringer Ingelheim Investigational Site, Killeen, Texas
  - 205.479.01038 Boehringer Ingelheim Investigational Site, Ettrick, Virginia
  - 205.479.01047 Boehringer Ingelheim Investigational Site, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this 12-week, randomised, double-blind, placebo-controlled, parallel group, multi-center Phase IV trial in chronic obstructive pulmonary disease (COPD), 140 patients were randomised to either Tiotropium 18 mcg or Placebo. Sixty eight (68) patients received Tiotropium 18 mcg and seventy two (72) patients received Placebo.
Groups:
- Placebo: placebo - Placebo Inhalation capsule, HandiHaler®
- Tiotropium 18 mcg: active - Tiotropium bromide Inhalation capsule 18 mcg, HandiHaler®
Period: Overall Study
Arm/Group | Placebo | Tiotropium 18 mcg
Started | 72 | 68
Completed | 68 | 66
Not Completed | 4 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Refused to continue medication | 2 | 1
Not completed — Due to other reason | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Tiotropium 18mcg: active - Tiotropium bromide Inhalation capsule 18 mcg, HandiHaler®
- Total: Total of all reporting groups
Arm/Group | Placebo | Tiotropium 18mcg | Total
Number analyzed (Participants) | 72 | 68 | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 59 | 53 | 112
  >=65 years | 13 | 15 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (8.7) | 59.2 (8.5) | 58.0 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 43 | 77
  Male | 38 | 25 | 63
Trough forced expiratory value (FEV1) [Mean (Standard Deviation); unit: Litre] | 1.75 (0.65) | 1.56 (0.61) | 1.65 (0.64)

OUTCOME MEASURES:

1. Primary Outcome: Trough FEV1 After 12 Weeks on Study Drug
Description: The primary endpoint was trough forced expiratory volume in 1 second (FEV1) after 12 weeks on study drug. Trough forced expiratory volume in 1 second (FEV1)was defined as the FEV1 measurement prior to the next dosing of study drug and approximately 24 hours after the last inhalation of study drug.
Time Frame: 12 weeks
Population: Treated Set (TS) with non missing FEV1 data.
Measure: Least Squares Mean (Standard Error); unit: Litre
Arm/Group | Placebo | Tiotropium 18 mcg
Number analyzed (Participants) | 67 | 67
Litre | 0.0378 (0.0383) | 0.0947 (0.0390)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium 18 mcg; Tiotropium 18 mcg minus Placebo; Test type: Superiority or Other; p = 0.3025, Mixed effect repeated measures (MMRM); Fixed effects:treatment,visit,treatment by visit,baseline and baseline by visit. Random:Patient. A spatial power covariance structure was used; Mean Difference (Final Values) = 0.0569, 95% CI 2-sided [-0.0516 to 0.1654], Standard Error of Mean 0.0550

2. Secondary Outcome: Time to Recovery From Acute Respiratory Symptoms
Description: Time to recovery was assessed with the EXACT-PRO questionnaire tool. The EXACT-PRO was designed to collect data to quantify frequency, severity, and duration of exacerbations in patients with COPD including the onset of and the recovery from COPD exacerbations.
  The EXACT-PRO is a 14-item questionnaire. Each attribute or item was assessed on a five- or six-point ordinal scale and summed to yield a total score that was converted to a 0-100 scale, with higher scores indicating a more severe health state or exacerbation.
  The EXACT-PRO was answered by the patients on a daily basis in the evening.
Time Frame: 12 weeks
Population: TS with non missing EXACT-PRO data.
Measure: Geometric Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Tiotropium 18 mcg
Number analyzed (Participants) | 70 | 67
units on a scale | 48.44 (12.33) | 47.86 (11.95)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium 18 mcg; Comparison Tiotropium 18 mcg Vs Placebo; Test type: Superiority or Other; p = 0.7823, 2sample t quantiles with pooled variance; Geometric mean ratio = 0.99, 95% CI 2-sided [0.9053 to 1.0780], Standard Error of Mean 0.44

3. Secondary Outcome: Trough FVC (in Litres) at 12 Weeks
Description: The trough Forced Vital Capacity (FVC) was defined as the FVC measurement prior to the next dosing of study drug and approximately 24 hours after the last inhalation of study drug.
Time Frame: 12 weeks
Population: TS with non missing FVC data.
Measure: Least Squares Mean (Standard Deviation); unit: Litres
Arm/Group | Placebo | Tiotropium 18 mcg
Number analyzed (Participants) | 67 | 67
Litres | 3.1537 (0.9772) | 2.9097 (0.9675)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium 18 mcg; Test type: Superiority or Other; p = 0.9025, Mixed effects repeated measures (MMRM) — Comparison Tiotropium 18 mcg Vs Placebo at Week 12; Fixed effects:treatment,visit,treatment by visit,baseline and baseline by visit. Patient was random. A spatial power covariance structure was used; Mean Difference (Final Values) = 0.0099, 95% CI 2-sided [-0.1489 to 0.1686], Standard Error of Mean 0.0806

4. Secondary Outcome: Responder Status at Week 4 Clinic Visit
Description: Responder status was determined at each clinic visit. The number and percentage of subjects in each of the following 3 classes were presented:
  * Subject recovered without change of therapy (subjects who received an additional course of antibiotics and/or systemic corticosteroids starting after Visit 1 were not included).
  * Subject recovered but had a change in therapy (subject received an additional course of antibiotics and/or systemic corticosteroids starting after Visit 1).
  * Subject did not recover.
Time Frame: 4 weeks
Population: Responder defined by >= 20% improvement. TS with non missing responder data.
Measure: Number; unit: participants
Arm/Group | Placebo | Tiotropium 18 mcg
Number analyzed (Participants) | 70 | 67
participants
  Week 4: Responder without therapy change | 38 | 39
  Week 4: Responder with changed therapy | 1 | 2
  Week 4: Non-responder | 31 | 26

5. Secondary Outcome: Responder Status at Week 12 Clinic Visit
Description: as for outcome 4
Time Frame: 12 weeks
Population: TS with non missing responder data at week 12. Responder defined by >= 20% improvement. .
Measure: Number; unit: participants
Arm/Group | Placebo | Tiotropium 18 mcg
Number analyzed (Participants) | 66 | 58
participants
  Week 12: Responder without therapy change | 34 | 34
  Week 12: Responder with changed therapy | 0 | 0
  Week 12: Non-responder | 32 | 24

6. Secondary Outcome: Weekly Rescue Medication Use Over the 12 Weeks of Study
Description: Daily rescue albuterol use was recorded in the diary in response to the following question: How many puffs of rescue medication did you use during the last 24 hours? The weekly rescue medication use was derived by summing the daily uses over the 12 weeks and dividing this total by 12 weeks.
Time Frame: 12 weeks
Population: TS with non missing rescue medication use.
Measure: Mean (Standard Deviation); unit: puffs
Arm/Group | Placebo | Tiotropium 18 mcg
Number analyzed (Participants) | 72 | 68
puffs | 17.0 (18.9) | 12.9 (16.6)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium 18 mcg; Comparison Tiotropium 18 mcg Vs Placebo Over 12 Weeks; Test type: Superiority or Other; p = 0.1797, t-test, 2 sided; 95% confidence interval is based on 2 sample t quantiles using pooled variance; Mean Difference (Final Values) = -4.0610, 95% CI 2-sided [-10.0157 to 1.8938], Standard Error of Mean 3.0115

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Placebo | Tiotropium 18 mcg
Serious Adverse Events (participants affected / at risk) | 3/72 | 3/68
Other Adverse Events (participants affected / at risk) | 8/72 | 6/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=72) | Tiotropium 18 mcg (N=68)
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=72) | Tiotropium 18 mcg (N=68)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 8 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.